CLINICAL TRIAL: NCT06609343
Title: Bupropion for Fatigue in End-stage Kidney Disease Patients on Hemodialysis (BRISK)
Brief Title: Bupropion for Fatigue in End-stage Kidney Disease Patients on Hemodialysis
Acronym: BRISK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Subrata Debnath, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000814
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease; Fatigue
Keywords: Hemodialysis; Kidney dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue | interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: A phase 2, open-label, single-arm, single-center, prospective, fixed-dose, 8-week intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hemodialysis Group (Experimental): Fixed dose bupropion hydrochloride 150 mg extended-release tablets will be administered orally thrice a week during routine dialysis sessions for consecutive 8 weeks.
  Interventions: Drug: Bupropion Hydrochloride 150 MG

INTERVENTIONS:
Drug: Bupropion Hydrochloride 150 MG — Bupropion Hydrochloride Extended Release is administered orally three times a week during routine dialysis sessions for 8 consecutive weeks

SUMMARY:
Fatigue is the most common symptom reported by end-stage kidney disease patients on maintenance hemodialysis. Unfortunately, there currently is no medical management for this overwhelming feeling of tiredness. As a result, patients continue to suffer with poor quality of life and impaired daily activities. The purpose of this pilot trial is to find out if bupropion (a medicine commonly prescribed for stopping smoking, seasonal mood disorder, and depression) may help lessen fatigue in hemodialysis patients.

In this study, hemodialysis participants will receive bupropion tablet orally three times a week during routine dialysis procedure for consecutive 8 weeks. Study participants will complete a battery of questionnaires to self-report fatigue, cognition, and quality of life. The study team will collect biological specimens. All these procedures will be performed at the dialysis clinic during routine dialysis procedure.

DETAILED DESCRIPTION:
While taking part in this study, participants will be asked to complete study procedures with the researchers or study staff three times a week during routine dialysis visits. Collections of blood, urine (if available) and stool will be collected at different time points over the 8-week intervention. Blood will be analyzed for markers of inflammation, amino acids, and for safety labs as needed. Blood will also be tested for pharmacokinetics of bupropion.

Primary Objective: To evaluate the feasibility and efficacy of bupropion for the treatment of fatigue in patients with end-stage kidney disease on maintenance hemodialysis.

Secondary Objective: To evaluate the effect of bupropion in reducing inflammatory markers in hemodialysis patients with fatigue.

Exploratory Objective: To examine whether bupropion improves cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ESKD patients between aged 25-74 yrs on maintenance in-center hemodialysis procedure 3 times/week for ≥3 months with an arteriovenous fistula or graft.
2. Blood hemoglobin of ≥10.0 g/dL based on most recent routine laboratory profile.
3. Dialysis adequacy measured with Kt/V of ≥1.2
4. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Currently on bupropion or hypersensitivity/ intolerance to bupropion by history and monoamine oxidase inhibitors.
2. Diagnosis or history of eating disorders (bulimia or anorexia nervosa) and seizure.
3. Pregnant, lactating, childbearing women
4. History of post-acute COVID-19 syndrome
5. Diagnosis of depression and/or on antidepressants and bipolar affective disorder
6. Patient Health Questionnaire (PHQ)-9 score of ≥10
7. Diagnosis of cognitive impairment including dementia
8. Current participation in another interventional trial
9. Scheduled for kidney transplantation in next 6 months
10. Life expectancy <6 months as judged by the attending nephrologist/primary care physician.
11. Current or history of substance abuse or dependency.

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Fatigue Inventory (BFI) Global Score | Baseline to 8 weeks
  This inventory contains 9 items scored from 0-10 with a total possible raw score of 0-90. A lower score indicates that there is less fatigue

SECONDARY OUTCOMES:
Change in plasma concentration of inflammatory marker IL-6 | Baseline to 8 weeks
  Plasma level of inflammatory marker of interleukin-6 (IL-6)
Change in plasma concentration of inflammatory marker TNF-α | Baseline to 8 weeks
  Plasma level of tumor necrosis factor-alpha (TNF-α)

OTHER OUTCOMES:
Change in Cognitive function using Trail Making Test B | Baseline to 8 weeks
  The participant will need a pencil to perform each part. The examiner starts timing as soon as the instructions are completed and the participant is signaled to begin. Timing is continued until the participant completes or discontinues the test. The time to completion in seconds is recorded. The maximum score for Part B is 300 seconds with 301" indicating the test was discontinued. A lower score indicates that the participant has better cognitive function and completed the task faster.
Change in Mini-COG score | Baseline to 8 weeks
  The score is made up of 2 parts: recall score is 0-3 points, 1 point is assigned for each word correctly recalled without prompt, so the score is higher if more words are recalled. For the clock drawing score, the possible score is 0-2 points, a higher score indicates more accuracy. The total score is between 0-5 with a higher score indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Subrata Debnath, MB.BS, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Hospital Dialysis Medical Center (DMC), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Any manuscript, abstract or other publication or presentation of results or information arising in connection with the trial (including any ancillary trial involving trial participants) must use deidentified data.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion at the time of publication in a peer review journal